CLINICAL TRIAL: NCT00156221
Title: MR Scanning of Very Young Children With Severe Developmental Disorders (Autistic Spectrum Disorders and/or Mental Retardation and/or Language Disorders)
Brief Title: MR Scanning of Very Young Children With Severe Developmental Disorders
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Collaborators: Netherlands Organisation for Scientific Research (Other Government); The Dutch Brain Foundation (Other)
Other Study IDs: METC UMC Utrecht 99/184
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2005-09

CONDITIONS: Autism; Mental Retardation; Language Disorder
Keywords: Autism; MRI; Developmental Disorders
MeSH Terms: conditions — Autistic Disorder; Intellectual Disability; Language Disorders; Developmental Disabilities

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Other

SUMMARY:
The specific is to study the MR morphologic and spectroscopic brain correlates and predictors of development in children with severe developmental disorders (autistic spectrum disorders and/or mental retardation and/or language disorders). Given the frequently observed association of autism with known medical conditions, particularly in cases with comorbid mental retardation and in cases with atypical autism (Rutter et al., 1994; Gillberg, 1995), children with suspected autism or related developmental disorders will be asked to participate in an extensive state of the art laboratory work-up which includes T1 and T2 weighted MRI of the brain. MRI data will be analyzed both qualitatively, looking for focal abnormalities and degree of myelination, and quantitatively, measuring volumes of total brain, cerebellum, ventricles and grey and white matter. For research purposes, the work-up will be supplied with proton Magnetic Resonance Spectroscopy (MRS) of the brain. This data set provides the opportunity to chart brain-behavior relationships in young children with suspected autism and related PDD cross-sectionally.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 months to 7 years
* Diagnosis of autism spectrum disorder, a language disorder or mental retardation

Exclusion Criteria:

* Significant motor or sensory impairment
* Major physical abnormalities
* History of serious head injury
* Identifiable neurologic disorder
* Metal implants
* Contraindication for MRI

Ages: 18 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2000-09; Study Completion 2005-09

CONTACTS AND LOCATIONS:
Overall Officials: Herman van Engeland, PhD, MD, Study Chair — UMC Utrecht; Mijke Zeegers, Msc, Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Netherlands